CLINICAL TRIAL: NCT03612648
Title: Evaluation of Three Fraction Accelerated Partial Breast Irradiation as the Sole Method of Radiation Therapy for Low-risk Stage 0 and I Breast Carcinoma
Brief Title: Three Fraction Accelerated Partial Breast Irradiation as the Sole Method of Radiation Therapy for Low-risk Stage 0 and I Breast Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201808046
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Breast Carcinoma; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TRI-APBI (Experimental): * Brachytherapy TRI-APBI the PTV is prescribed 7.5 Gy x three fractions given over two to three days OR
  * External beam TRI-APBI the PTV is prescribed 8.5 Gy x three fractions given over two to three days
  Interventions: Radiation: Three Fraction Accelerated Partial Breast Irradiation; Procedure: Partial mastectomy

INTERVENTIONS:
Radiation: Three Fraction Accelerated Partial Breast Irradiation — * TRI-APBI simulation must take place no more than 8 weeks from final definitive breast surgery
  * Machines that could be used include: SAVI applicator, The ViewRay System for Radiation Therapy, The ViewRay (MRIdian) Linac System, Halcyon, True Beam, True Beam STx, Edge Radiotherapy Delivery System
  Other Names: TRI-APBI
Procedure: Partial mastectomy — -Standard of Care

SUMMARY:
The investigators proposed approach allows them to deliver a low total dose of radiation to patients with low-risk, early-stage breast cancer which would further minimize the impact of adjuvant therapy. This work has the potential to revolutionize partial breast irradiation by allowing it to take place at many radiation oncology centers with minimal specialized equipment beyond that commonly available. The investigators first step is this proposed single institution phase I/II study designed primarily to evaluate the tolerance of this approach which the investigators are choosing to call Three Fraction APBI (Tri-APBI).

ELIGIBILITY:
Inclusion Criteria:

* AJCC 7th Edition stage 0 or I (TisN0 ≤ 2 cm or T1N0) histologically confirmed carcinoma of the breast, treated with partial mastectomy. Axillary sampling is required only for cases of invasive cancers. Tumor size is determined by the pathologist. Clinical size may be used if the pathologic size is indeterminate. Patients with invasive cancer must have no positive axillary lymph nodes with at least 6 axillary lymph nodes sampled or a negative sentinel node.
* Negative histologic margins of partial mastectomy or re-excision specimen. Margins generally are positive if there is invasive or noninvasive tumor at the inked resection margin, close but negative if the tumor is within 2 mm of the inked margin and negative if the tumor is at least 2 mm away from the inked edge.
* Invasive ductal, lobular, medullary, papillary, colloid (mucinous), tubular histologies, or mixed histologies (lesions ≤ 2 cm) that are estrogen or progesterone receptor positive and do not exhibit HER2/neu gene amplification OR ductal carcinoma in situ (lesions ≤ 2 cm).
* Neoadjuvant hormone therapy, chemotherapy, or biologic therapy is not allowed prior to TRI-APBI, but adjuvant hormone therapy may have been started after surgery. Planned chemotherapy or biologic therapy must not start for at least 4 weeks after the completion of TRI-APBI.
* Good candidate for treatment per protocol in the judgment of the PI and/or treating physician following simulation.
* Postmenopausal status.
* Age ≥ 50 years at diagnosis.
* Able to understand and willing to sign IRB-approved written informed consent document.
* English speaker.
* All radiation therapy must be planned for delivery at BJH. External beam patients will be treated at BJH on a Viewray Unit, the Varian Edge unit, or the Varian Halcyon unit. Brachytherapy cases will be treated in the BJH brachytherapy center. Pre and post treatment care is allowed at any Siteman center.

Exclusion Criteria:

* Presence of distant metastases.
* Nonepithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (tumors in different quadrants of the breast, or tumors separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
* Histologically confirmed positive axillary nodes in the ipsilateral axilla. Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy or chemotherapy.
* Diagnosis of systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Diagnosis of a coexisting medical condition which limits life expectancy to < 2 years.
* History of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Paget's disease of the nipple.
* Skin involvement, regardless of tumor size.
* Unsatisfactory breast for TRI-APBI as determined by the treating physician. For example, if there is little breast tissue remaining between the skin and pectoralis muscle after surgery, treatment with TRI-APBI is technically problematic.
* Partial mastectomy so extensive that the cosmetic result is fair or poor prior to TRI-APBI as determined by the treating physician.
* Surgical margins which cannot be microscopically assessed or are positive at pathological evaluation.
* Time between final definitive breast procedures to TRI-APBI simulation is greater than 8 weeks.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Tolerance of Tri-APBI as measured by the rate of acute treatment-related grade 3 or higher toxicity or any other grade 4 or 5 toxicity attributed to treatment | Through 8 weeks
  * Adverse events will be graded using CTCAE Version 5.0
  * Toxicities of concern include breast pain, delayed wound healing, persistent seroma fluid accumulation, breast fibrosis, and fat necrosis in the treated breast. Rare toxicities include radiation pneumonitis, coronary artery disease, and pericarditis
Ipsilateral breast tumor recurrence rate | 5 years after treatment
  -Recurrence of breast cancer in the treated breast is an ipsilateral breast tumor recurrence (IBTR)
Tolerance of Tri-APBI as measured by the rate of late treatment-related grade 3 or higher toxicity or any other grade 4 or 5 toxicity attributed to treatment | Through 5 years after treatment
  * Adverse events will be graded using CTCAE Version 5.0
  * Toxicities of concern include breast pain, delayed wound healing, persistent seroma fluid accumulation, breast fibrosis, and fat necrosis in the treated breast. Rare toxicities include radiation pneumonitis, coronary artery disease, and pericarditis

SECONDARY OUTCOMES:
Proportion of participants who are free of breast cancer recurrence in the regional lymph nodes | 5 years after treatment
  -Defined as ipsilateral axilla, infraclavicular, supraclavicular, and internal mammary groups
Proportion of participants who are free of breast cancer distant metastases | 5 years after treatment
Change in Quality of life as measured by the EORTC QLQ-30 questionnaire | Through 5 years after treatment
  The QLQ-C30 includes 6 general questions and 24 questions in 9 subscales measuring physical, role, emotional, cognitive and social function, as well as global health status, nausea/ vomiting, pain and fatigue
  * Each of the subscales will be tabulated and presented graphically over the assessment times. Mixed repeated measures models will be generated to describe the nature of change in quality of life over time
  * Responses vary from 1=Not at All to 4 = Very Much
Change in Quality of life as measured by the EORTC QLQ-BR23 questionnaire | Through 5 years after treatment
  * The QLQ-B23 provides 23 questions in 8 breast cancer specific subscales, 4 measuring symptoms and 4 measuring function
  * Each of the subscales will be tabulated and presented graphically over the assessment times. Mixed repeated measures models will be generated to describe the nature of change in quality of life over time
  * Responses vary from 1=Not at All to 4 = Very Much
Change in Cosmesis as measured by the Breast Retraction Assessment | Through 5 years after treatment
  * Cosmesis will be graded by the patient and the radiation oncologist (or nurse practitioner) before treatment, 6-10 weeks after TRI-APBI, at 4-8 month follow-up, at 10-14 month follow-up, and at yearly intervals thereafter for a total of 5 years following TRI-APBI
  * The Breast Retraction Assessment consists of measuring certain parts of a participant's chest and then using a formula to come up with the measurements
Change in Cosmesis as measured by the Percent Breast Retraction Assessment | Through 5 years after treatment
  * Cosmesis will be graded by the patient and the radiation oncologist (or nurse practitioner) before treatment, 6-10 weeks after TRI-APBI, at 4-8 month follow-up, at 10-14 month follow-up, and at yearly intervals thereafter for a total of 5 years following TRI-APBI
  * The Percent Breast Retraction Assessment consists of measuring certain parts of a participant's chest and then using a formula to come up with the measurements
Change in Cosmesis as measured by the Aronson modified Harris scale | Through 5 years after treatment
  * Cosmesis will be graded by the patient & radiation oncologist (or nurse practitioner) before treatment, 6-10 weeks after TRI-APBI, 4-8 month follow-up, 10-14 month follow-up, & yearly intervals for a total of 5 years following TRI-APBI
  * The Aaronson modification of the Harris scale will be used to evaluate cosmesis & the scale consists of:
    * Excellent-when compared to the untreated breast, there is minimal or no difference in the size, shape or texture of the treated breast - may be mild thickening or scar tissue within the breast or skin, but not enough to change the appearance
    * Good-mild asymmetry in the size or shape of the treated breast as compared to the normal breast. The thickening or scar tissue within the breast causes only a mild change in the shape
    * Fair-obvious difference in the size & shape of the treated breast. This change involves 1/4 or less of the breast
    * Poor-marked change in the appearance of the treated breast involving more than 1/4 of the breast tissue
Presence of complications using CTCAE Version 5.0 criteria | Through 5 years after treatment
Proportion of participants undergoing mastectomy on the treated side | 5 years after treatment
Frequency of any CTCAE Version 5.0 grade 3-4 toxicities | Through 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu